CLINICAL TRIAL: NCT03024619
Title: A Pilot Study of the Correlation Between Symptoms of Interstitial Cystitis and Urinary pH
Brief Title: Interstitial Cystitis and Urinary pH
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Iona Marcu, MD, Principal Investigator, St. Louis University
Other Study IDs: 26300
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pain and Urinary pH — assess the correlation between urinary pH and Interstitial Cystitis (IC) pain, with emphasis placed on exploring the type and severity of pain

SUMMARY:
This is a pilot study to assess the correlation between urinary pH and Interstitial Cystitis (IC) pain, with emphasis placed on exploring the type and severity of pain.

DETAILED DESCRIPTION:
Subjects who agree to participate in the study will meet with a research team member who will review the study with them, obtain informed consent sign the HIPPA form, and provide study materials (void diary for urine quantification and recording of IC symptoms, pH strips to dip urine, "hat" to measure urine). Medical charts will be reviewed to determined how Interstitial Cystitis was diagnosed, medications, medical/surgical history, and demographics such as weight, height, BMI, race, age, marital status, education, insurance, tobacco or alcohol use. Subjects will need to dip pH paper into the urine and specific gravity reagent strip, and, by color comparison between the strips and the corresponding scales, determine and record urine pH and specific gravity. They will need to fill out the corresponding section in the voiding diary that is a survey to type and severity or pain as well as other symptoms of IC. The research team member will teach the subject how to measure the volume of their urine and how to measure and record specific gravity and pH. When not practical to record the volume of the urine (when patients are at work or away from home) they will still be asked to record pH, specific gravity and experienced symptoms. Subjects will be asked to perform the above described protocol with each episode of micturition for 3 days.

After enrollment, subjects will complete the O'Leary-Sant pain (symptom and problem index) questionnaire, if subjects have a combined score greater than or equal to 12 they are considered to have problematic or symptomatic IC. The voiding diary that include pH and specific gravity measurement measurements, times, volume, and survey of symptoms will be returned 1-2 weeks following completion of 3 day void diary for a face-to-face meeting with a research team member. Attempts will be made to have those meetings coincide with a clinical visit to minimize study burden to the subject(e.g. - at the time of cystoscopy or follow-up visit. )

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70, with diagnosed Interstitial Cystitis (IC) and bladder pain present during week preceding enrollment.

Exclusion Criteria:

* Subjects who are pregnant. Subjects with current UTI or are unwilling/unable to provide consent.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with symptomatic diagnosed Interstitial Cystitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Correlation between urinary pH and bladder pain. | 3 days
  Measure urine pH and visual analog pain scale score and describe correlation between them.

SECONDARY OUTCOMES:
Correlation between urinary specific gravity and bladder pain. | 3 days
  Measure urine specific gravity and visual analog pain scale score and describe correlation between them.

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Marcu, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No